CLINICAL TRIAL: NCT01530321
Title: Dose-Response of Manipulation for Cervicogenic Headache
Brief Title: Cervicogenic Headache Dose-Response
Acronym: CGH D-R
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Western States (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Mitchell Haas, Associate Vice President of Research, University of Western States
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R01AT006330 (NIH)
Record Dates: First submitted 2012-02-02; First posted 2012-02-09 (Estimated); Last update posted 2018-11-20 (Actual); Status verified 2018-11

CONDITIONS: Cervicogenic Headache
Keywords: cervicogenic headache; spinal manipulation; chiropractic; randomized controlled trial; dose-response; efficacy
MeSH Terms: conditions — Post-Traumatic Headache | interventions — Manipulation, Spinal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- High dose spinal manipulation (Experimental): 18 visits for spinal manipulation
  Interventions: Other: Spinal Manipulation
- Moderate dose spinal manipulation (Experimental): 12 visits for spinal manipulation and 6 visits for light massage
  Interventions: Other: Spinal Manipulation; Other: Light Massage
- Low dose spinal manipulation (Experimental): 6 visits for spinal manipulation and 12 visits for light massage
  Interventions: Other: Spinal Manipulation; Other: Light Massage
- High dose massage (Other): 18 visits for light massage
  Interventions: Other: Light Massage

INTERVENTIONS:
Other: Spinal Manipulation — 5 minutes of high velocity, low amplitude thrust to cervical and upper thoracic spine.
  Arms: High dose spinal manipulation; Low dose spinal manipulation; Moderate dose spinal manipulation
Other: Light Massage — 5 minutes of light pressure massage to the neck and upper back
  Arms: High dose massage; Low dose spinal manipulation; Moderate dose spinal manipulation

SUMMARY:
This study will determine the number of visits to a chiropractor for spinal manipulation and light massage necessary for the optimal relief of cervicogenic headache (headache with associated neck pain). Effectiveness of care will also be determined.

ELIGIBILITY:
Inclusion Criteria:

* chronic cervicogenic headache
* threshold pain level
* threshold headache frequency
* independently ambulatory
* English literate
* candidate for spinal manipulation

Exclusion Criteria:

* contraindication to thrust spinal manipulation or massage
* most other headache types
* Recent manual/exercise therapy from licensed provider for head/neck
* threshold pain medication use
* pregnancy
* involvement with another pain study
* suspicion of unmanaged depression
* most cancers
* hypertension (at least stage II)
* complicating neurological/spinal conditions
* pre-randomization noncompliance or cannot/will not comply with protocols
* health-related litigation, claims, or disability compensation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 256 (Actual)
Dates: Start 2012-08; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Headache days change from baseline for cervicogenic headache | 0, 6, 12, 24, 39, 52 weeks
  Days with cervicogenic headache in the last four weeks from a daily headache diary. Change score = follow-up score - baseline score)

SECONDARY OUTCOMES:
Average pain change from baseline for cervicogenic headache | 0, 6, 12, 24, 39, 52 weeks
  Average cervicogenic headache pain in the last four weeks evaluated by averaging daily headache diary pain scores. Pain is rated on a 0 to 11 numeric rating scale.
Headache-related disability change from baseline for cervicogenic headaches | 0, 6, 12, 24, 39, 52 weeks
  Headache Impact Test (HIT-6)
Headache-related disability days change from baseline | 0, 6, 12, 24, 39, 52 weeks
  Number of days in the last four weeks from recall unable to carry out daily work for at least one half day because of cervicogenic headache.
EuroQol-5D change from baseline | 0, 12, 24, 39, 52 weeks
  Health-related quality of life
Average pain change from baseline for neck | 0, 6, 12, 24, 39, 52 weeks
  Average neck pain in the last four weeks from recall. Pain is rated on a 0 to 11 numeric rating scale.
Neck pain days change from baseline | 0, 6, 12, 24, 39, 52 weeks
  Number of days with neck pain in last 4 weeks from recall.
medication use change from baseline | 0, 6, 12, 24, 39, 52 weeks
  Number days of use of prescription and nonprescription medications for headaches with neck pain
Outside Care change from baseline | 0, 6, 12, 24, 39, 52 weeks
  Visits to providers outside the study for care of cervicogenic headache. Includes hospital and emergency room visits
Patient Satisfaction | week 12
  Likert scale for success of care
Objective biomechanical measures change from baseline | 0, 6 weeks
  Measures of cervical joint function and kinematics including global range of motion, spinal segmental joint restriction, pain pressure thresholds
Quality-adjusted life years change from baseline | 0, 12, 24, 39, 52 weeks
  utility for cost-effectiveness analysis
Direct & Indirect costs change from baseline | 0, 6, 12, 24, 39, 52 weeks
  Health services; lost work days and productivity
Perceived headache average pain change from baseline for cervicogenic headache | 0, 6, 12, 24, 39, 52 weeks
  Perceived change in average pain from baseline on a -10 to +10 (21-point) numeric rating scale
Perceived headache improvement from baseline for cervicogenic headache | 0, 6, 12, 24, 39, 52 weeks
  Perceived cervicogenic headache improvement from baseline on a 9-point Likert-like scale.

CONTACTS AND LOCATIONS:
Overall Officials: Mitchell Haas, DC, MA, Principal Investigator — University of Western States; Gert Bronfort, DC, PhD, Principal Investigator — University of Minnesota
Locations (2):
- United States (2):
  - Northwestern Health Sciences University, Bloomington, Minnesota
  - University of Western States, Portland, Oregon

REFERENCES:
- [Background] Hanson L, Haas M, Bronfort G, Vavrek D, Schulz C, Leininger B, Evans R, Takaki L, Neradilek M. Dose-response of spinal manipulation for cervicogenic headache: study protocol for a randomized controlled trial. Chiropr Man Therap. 2016 Jun 8;24:23. doi: 10.1186/s12998-016-0105-z. eCollection 2016. PMID 27280016
- [Result] Haas M, Bronfort G, Evans R, Schulz C, Vavrek D, Takaki L, Hanson L, Leininger B, Neradilek MB. Dose-response and efficacy of spinal manipulation for care of cervicogenic headache: a dual-center randomized controlled trial. Spine J. 2018 Oct;18(10):1741-1754. doi: 10.1016/j.spinee.2018.02.019. Epub 2018 Feb 23. PMID 29481979